CLINICAL TRIAL: NCT05029063
Title: Primary Thromboprophylaxis in Patients With Malignancy and Central Venous Catheters: a Randomized Controlled Trial
Brief Title: Primary Thromboprophylaxis in Patients With Malignancy and Central Venous Catheters
Acronym: TRIM-Line
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TRIM-Line 3698
Record Dates: First submitted 2021-06-30; First posted 2021-08-31 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Venous Thromboembolism; Cancer
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Rivaroxaban 10mg OD
  Interventions: Drug: Rivaroxaban 10 MG
- Control (Placebo Comparator): Identical Placebo 10mg OD
  Interventions: Drug: Rivaroxaban 10 MG

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Identical comparator drug
  Other Names: Placebo

SUMMARY:
The purpose of the full trial is to determine the efficacy and safety of prophylactic dose rivaroxaban to prevent VTE among cancer patients with CVC.

DETAILED DESCRIPTION:
TRIM-Line is a double blind randomized controlled trial comparing rivaroxaban 10mg po daily vs placebo in patients with active cancer and indwelling CVC. This will involve 9 centers across Canada.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with a new or existing diagnosis of cancer and a CVC inserted in the last 72 hours.

Exclusion criteria:

1. CVC in place for >72 hours
2. Patient requires anticoagulation for other indications
3. Concomitant use of dual antiplatelet therapy
4. Major bleeding event in the last 4 weeks
5. Patients receiving concomitant systemic treatment with strong inhibitors of both CYP 3A4 and P-gp (such as cobicistat, ketoconazole, itraconazole, posaconazole, or ritonavir).
6. Known pregnancy or plan to become pregnant in next 3 months
7. Severe renal insufficiency (Creatinine clearance <30 mL/min (defined by Cockcroft-Gault) in the previous 3 months
8. Documented severe liver disease (e.g., acute clinical hepatitis, chronic active hepatitis or cirrhosis) in the previous 3 months
9. Known thrombocytopenia (platelet count < 50x 109/L) in the previous 3 months
10. Known allergy to rivaroxaban
11. Life expectancy <3 months
12. History of condition at increased bleeding risk including, but not limited to:

    1. cerebral infarction (hemorrhagic or ischemic), active peptic ulcer disease with recent bleeding, spontaneous or acquired impairment of hemostasis in the past 4 weeks.
    2. Chronic hemorrhagic disorder
13. Primary malignancy diagnosis of basal cell or squamous cell carcinoma of the skin only
14. Refused or unable to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1828 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Major VTE prevention | 90 days (± 3 days) of randomization
  Number of Major VTE's in patient population
Episodes of Major Bleeding | 90 days (± 3 days) of randomization
  Number of participants who had a major bleed

SECONDARY OUTCOMES:
Number of participants with Clinically Relevant Non-Major Bleeding (CRNMB) | 90 days (± 3 days) of randomization
  As defined by ISTH
Number of patients who had a fatal VTE | 90 days (± 3 days) of randomization
  Fatal VTE
Number of patients who benefitted from using the experimental intervention | 90 days (± 3 days) of randomization
  Composite of major VTE and major bleeding
PE | 90 days (± 3 days) of randomization
  Incidental and Symptomatic
Proximal CVC VTE | 90 days (± 3 days) of randomization
  Incidental and symptomatic proximal (axillary vein or more proximal) upper extremity CVC-related DVT
Distal CVC VTE | 90 days (± 3 days) of randomization
  Incidental and symptomatic distal (brachial vein) or proximal (axillary vein or more proximal) upper extremity CVC-related DVT
Proximal Lower extremity DVT | 90 days (± 3 days) of randomization
  Incidental and symptomatic proximal (popliteal vein or more proximal) lower extremity DVT
Distal Lower extremity DVT | 90 days (± 3 days) of randomization
  Incidental and symptomatic distal or proximal (popliteal vein or more proximal) lower extremity DVT
Number of participants with Unusual site thrombosis including: splanchnic vein (portal, splenic, superior mesenteric, inferior mesenteric, hepatic) cerebral vein, renal or gonadal vein thromboses | 90 days (± 3 days) of randomization
  Unusual site thrombosis including: splanchnic vein (portal, splenic, superior mesenteric, inferior mesenteric, hepatic) cerebral vein, renal or gonadal vein thromboses
Number of participants with Superficial upper or lower extremity vein thrombosis | 90 days (± 3 days) of randomization
  Superficial upper or lower extremity vein thrombosis
Number of participants with an arterial thromboembolic event including: MI, stroke, peripheral arterial disease | 90 days (± 3 days) of randomization
  Arterial thromboembolic events defined as a diagnostically confirmed final clinical diagnosis of myocardial infarction, stroke or peripheral arterial disease involving the following arterial vascular beds: carotid, upper or lower extremity, gastrointestinal tract, liver, spleen, or kidney
CVC Life-span | 90 days (± 3 days) of randomization
  Life span of inserted CVC
Number of patients with CVC occlusion occurring after the start of therapy, defined as an obstruction of the CVC lumen that prevents or limits the ability to flush, withdraw blood and/or administer solutions or medications. | 90 days (± 3 days) of randomization
  CVC occlusion occurring after the start of therapy, defined as an obstruction of the CVC lumen that prevents or limits the ability to flush, withdraw blood and/or administer solutions or medications.
Number of patients with CVC-related blood stream infection defined as the presence of bacteremia originating from the CVC according to the definition from the Centers for Disease Control and Prevention | 90 days (± 3 days) of randomization
  CVC-related blood stream infection defined as the presence of bacteremia originating from the CVC according to the definition from the Centers for Disease Control and Prevention
Number of participants who passed away during the trial | 90 days (± 3 days) of randomization
  Overall mortality
EQ-5D-5L Health-related quality of life | 90 days (± 3 days) of randomization
  Health-related quality of life
ICER | 1 Year
  Incremental cost-effectiveness ratio (ICER) at one year

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Marc Carrier, Principal Investigator — Ottawa Hospital Research Institute
Locations (11):
- Canada (11):
  - Nova Scotia Health, Halifax, Nova Scotia
  - William Osler Health System, Brampton, Ontario
  - HHS - Juravinski Hospital, Hamilton, Ontario
  - Ottawa Hospital Research Institute- The Ottawa Hospital, Ottawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Niagara Health, St. Catharines, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - CISSS Montérégie-Centre HOPITAL CHARLES LEMOYNE, Greenfield Park, Quebec
  - Centre Intégré de santé et de services sociaux de Chaudière-Appalaches, Lévis, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikesaka R, Siegal D, Mallick R, Wang TF, Witham D, Webb C, Carrier M; Canadian Venous Thromboembolism Research Network (CanVECTOR). Thromboprophylaxis with rivaroxaban in patients with malignancy and central venous lines (TRIM-Line): A two-center open-label pilot randomized controlled trial. Res Pract Thromb Haemost. 2021 May 5;5(4):e12517. doi: 10.1002/rth2.12517. eCollection 2021 May. PMID 34027291